CLINICAL TRIAL: NCT00071968
Title: An Open-Label Study Of Exploratory Pharmacogenomics And Pharmacologic Effects Of Neoadjuvant Oral CCI-779 In Newly Diagnosed Prostate Cancer Patients Undergoing Radical Prostatectomy Who Have A High Risk Of Relapse
Brief Title: Neoadjuvant CCI-779 Followed By Radical Prostatectomy in Treating Patients With Newly Diagnosed Prostate Cancer Who Have a High Risk of Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000331979; UCLA-0306091; WYETH-C-3066A1-132-US
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer; stage I prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — temsirolimus; Neoadjuvant Therapy

INTERVENTIONS:
Drug: temsirolimus
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as CCI-779, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving CCI-779 before surgery may shrink the tumor so that it can be removed.

PURPOSE: This randomized phase II trial is studying how well CCI-779 works in treating patients who are undergoing radical prostatectomy for newly diagnosed prostate cancer at high risk of relapse.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effects of oral CCI-779 on changes in the phosphorylation state of proteins in the mammalian target of rapamycin (mTOR) signaling pathway in the tumor tissue of patients with newly diagnosed prostate cancer undergoing radical prostatectomy.
* Determine the effects of this drug on changes in p70S6 kinase activity, phosphorylation state of mTOR pathway proteins, and on global and targeted gene expression patterns in the peripheral blood mononuclear cells (PBMCs) of these patients.

Secondary

* Determine the effects of this drug on global and targeted gene expression patterns in these patients.
* Identify pharmacodynamic/pharmacogenomic surrogate markers of this drug in both tumor tissue and PBMCs and determine if blood may be used as a surrogate tissue source for biomarkers of drug activity in the tumor in these patients.
* Determine, preliminarily, the potential antitumor effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Correlate phosphatase and tensin homolog (PTEN) gene status with the pharmacodynamic/pharmacogenomic effects of this drug in these patients.
* Determine the effects of this drug on changes in protein expression patterns in the plasma of these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are randomized to 1 of 3 treatment arms. Patients randomized to arm III are stratified according to tumor expression of phosphatase and tensin homolog (PTEN) gene mutations (negative vs positive).

* Arm I: Patients receive oral CCI-779 once daily for a total of 8 weeks.
* Arm II: Patients receive a higher dose of CCI-779 as in arm I.
* Arm III: Patients receive a higher dose (higher than arm II) of CCI-779 as in arm I.

Approximately 24-48 hours after the last dose of CCI-779, patients in all arms undergo radical prostatectomy.

Patients are followed on day 7-10 and then at 4 weeks after study completion.

PROJECTED ACCRUAL: A total of 40 patients (5 each for arms I and II and 30 for arm III) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Diagnosis based on a minimum of 6 core biopsy samples
  * Clinically confirmed organ-confined disease
* Candidate for radical prostatectomy
* No evidence of metastatic disease by CT scan and bone scan
* High risk of relapse based on either of the following criteria:

  * Any one of the following:

    * Stage T2C or higher
    * Gleason score greater than 7
    * Prostate-specific antigen (PSA) greater than 20 ng/mL OR
  * Any two of the following:

    * Gleason score at least 7
    * PSA 10-20 ng/mL
    * Greater than 50% of total biopsy cores with cancer involvement

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* No active bleeding
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* No acute or chronic hepatitis B

  * Hepatitis B surface antigen negative
* No acute or chronic hepatitis C

  * No antibodies to hepatitis C
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2 times ULN

Renal

* No ongoing urinary tract infection necessitating rapid or emergent surgical resection
* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No unstable angina
* No myocardial infarction within the past 6 months
* No life-threatening ventricular arrhythmia requiring ongoing maintenance therapy

Pulmonary

* No known pulmonary hypertension
* No pneumonitis

Other

* Fertile patients must use effective contraception during and for 12 weeks after study participation
* HIV negative
* No other severe immunocompromised states
* No active infection requiring antibiotic therapy
* No serious concurrent illness
* No other major illness that would substantially increase the risk associated with study participation
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* More than 3 weeks since prior IV corticosteroids
* No concurrent systemic corticosteroids
* No prior or concurrent hormonal therapy for underlying malignancy

Radiotherapy

* No prior or concurrent radiotherapy

Surgery

* More than 3 months since prior major surgery

Other

* More than 1 month since prior experimental drugs
* More than 3 weeks since prior immunosuppressive agents
* No concurrent immunosuppressive therapies
* No other concurrent investigational agents
* No concurrent enzyme-inducing anticonvulsants (e.g., phenobarbital, phenytoin, or carbamazepine)
* No concurrent ketoconazole, diltiazem, rifampin, terfenadine, cisapride, astemizole, pimozide, or Hypericum perforatum (St. John's wort)
* No concurrent grapefruit or grapefruit juice

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-08; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Phosphorylation state of proteins
p70S6 kinase activity
Phosphorylation state of mTOR pathway proteins
Global and targeted gene expression patterns in peripheral blood mononuclear cells

SECONDARY OUTCOMES:
Global and targeted gene expression patterns
Pharmacodynamics and pharmacogenomic surrogate markers
Antitumor effects
Pharmacokinetics
Correlation of phosphatase and tensin homolog gene status with pharmacodynamic and pharmacogenomic effects
Protein expression patterns in the plasma

CONTACTS AND LOCATIONS:
Overall Officials: Charles Sawyers, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Thomas G, Speicher L, Reiter R, et al.: Demonstration that temsirolimus preferentially inhibits the mTOR pathway in the tumors of prostate cancer patients with PTEN deficiencies. [Abstract] Clin Cancer Res 11 (Suppl 24): A-C131, 2005.